CLINICAL TRIAL: NCT03374371
Title: Identification of Genomic Markers Associated With the Invasiveness of Staphylococcus Epidermidis Strains Responsible for Infections
Brief Title: Invasive Markers of Staphylococcus Epidermidis
Acronym: SepiNGS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI17029J; 2017-A02742-51 (Other: ID-RCB)
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Staphylococcus Epidermidis Positive Blood Culture
Keywords: Staphylococcus epidermidis Infection; Staphylococcus epidermidis Contamination; intravascular device; implanted material

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- S. epidermidis Infection (CASE): Patients with confirmed infection at S. epidermidis
  Interventions: Diagnostic Test: high-throughput sequencing
- S. epidermidis Contamination (CONTROL): Patients with confirmed contamination at S. epidermidis
  Interventions: Diagnostic Test: high-throughput sequencing

INTERVENTIONS:
Diagnostic Test: high-throughput sequencing — technique of high-throughput sequencing of the markers present in the genome of the S. epidermidis strains responsible for infection in order to help to discriminate the true infections of the contaminations

SUMMARY:
The purpose of the study is to identify biomarkers allowing the distinction between invasive and non-invasive strains of Staphylococcus epidermidis. This distinction is important to determine if the patient is infected and, as a consequence, if an antibiotic treatment is required.

DETAILED DESCRIPTION:
In the hospital, a large proportion of bacteraemia and implantable medical device infections are caused by Staphylococcus epidermidis. This microorganism is the most abundant on human skin and all patients are carriers. Its remarkable ability to form biofilms on most materials explains that catheter-related infections are by far the most common.

S. epidermidis infections are difficult to treat because most strains are multi-resistant and antibiotics are less effective in the presence of biofilms.

In addition, S. epidermidis poses a major diagnostic problem because it is also the first source of contamination of blood culture sample and intraoperative samples (in case of suspected infection of orthopedic material in particular). Thus, when a sample is positive for S. epidermidis, there is less than a 25% chance that it reflects true bacteremia in the patient and 30% of patients would inappropriately receive vancomycin following contaminated blood cultures. Differentiating a contamination of a blood or intraoperative sample from true S. epidermidis infection is therefore crucial for patient management because unnecessary antibiotic therapy is potentially responsible for the emergence of resistant strains, toxicity and additional costs.

The objective of this study is to identify the genetic markers that make it possible to differentiate the strains causing infections from the strains causing contamination by comparing their genomes using high throughput sequencing.

ELIGIBILITY:
Inclusion Criteria:

CASE Inclusion Criteria:

Population 1: nosocomial bacteraemia associated with intravascular devices

1. Hospitalized patient with intravascular device (peripheral or central, venous or arterial, short or long duration) for at least 48 hours before the development of bacteraemia
2. Presenting a definite infection with S. epidermidis according to the categorization criteria,

Sub-Population 1A:

3a) Aged less than 28 days (New-born)

Sub-population 1B:

3b) Aged 28 days or more

Population 2: nosocomial infections of implanted material

1. An operated patient carrying implanted equipment following orthopaedic surgery, following cardiac surgery or following neurosurgery,
2. Presenting a definite infection with S. epidermidis according to the categorization criteria occurring in the year following surgery

CONTROL Inclusion Criteria:

Population 1: carrier of intravascular devices

1. Hospitalized patient with intravascular device (peripheral or central, venous or arterial, short or long duration) for at least 48 hours before positive blood culture with S. epidermidis
2. Certain contamination with S. epidermidis according to the categorization criteria,

Sub-Population 1A:

3a) Aged less than 28 days (Newborn)

Sub-population 1B:

3b) Aged 28 days or more

Population 2: carrier of implanted material

1. An operated patient carrying implanted equipment following orthopedic surgery, following cardiac surgery or following neurosurgery,
2. Presenting a certain contamination to S. epidermidis according to the categorization criteria occurring in the year following surgery

Exclusion Criteria:

CASE Exclusion Criteria Population 1: nosocomial bacteremia associated with intravascular devices

1. Opposition of the patient or the holders of parental authority (minor patients)
2. Patient with polymicrobial infection
3. Patient with a colonized catheter (positive catheter end culture <103UFC / mL) with no clinical signs of local or general infection and with sterile peripheral blood cultures
4. Patient with local catheter infection (positive catheter end culture> 103UFC / mL) with local inflammatory signs only and with sterile peripheral blood cultures

Population 2: nosocomial infections of implanted material

1. Opposition of the patient or the holders of parental authority (minor patients)
2. Patient with an infection of material concomitant with a catheter-related infection

CONTROL Exclusion Criteria

Populations 1 and 2:

Opposition of the patient or the holders of parental authority (minor patients)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population 1 (bacteraemia related to intravascular devices) : patients hospitalized for at least 48 hours including new-borns
  Population 2 (infections of materials) : patients carrying medical devices implanted following an act of surgery (orthopedic, cardiac or neurosurgery)
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
genetic markers of S. epidermidis | at the time of the positive sampling of S. epidermidis
  to identify genetic markers associated with a significant risk of invasive S. epidermidis infections

SECONDARY OUTCOMES:
Correlation of the genotype with the characteristics of the infections | at the time of the positive sampling of S. epidermidis
  identification of genetic markers specifically associated with a type of infection (catheter-related bacteremia in newborns, catheter-related bacteremia in patients 28 days or older, infections of orthopedic equipment or infections of cardiac equipment)
Intra-hospital cross-transmission detection | at the time of the positive sampling of S. Epidermidis
  The comparison of the strains will be based on the study of the variations in the part of the genome that is common to all the strains to detect possible transfers between patients

CONTACTS AND LOCATIONS:
Overall Officials: Anne JAMET, MD, Principal Investigator — Assistance Public Hôpitaux de Paris (APHP)
Locations (1):
- Hôpital Necker Enfants Malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jamet A, Guglielmini J, Brancotte B, Coureuil M, Euphrasie D, Meyer J, Roux J, Barnier JP, Bille E, Ferroni A, Magny JF, Bole-Feysot C, Charbit A, Nassif X, Brisse S. High-Resolution Typing of Staphylococcus epidermidis Based on Core Genome Multilocus Sequence Typing To Investigate the Hospital Spread of Multidrug-Resistant Clones. J Clin Microbiol. 2021 Feb 18;59(3):e02454-20. doi: 10.1128/JCM.02454-20. Print 2021 Feb 18. PMID 33328176